CLINICAL TRIAL: NCT04548128
Title: Implantation of the HeartMate 3 in Subjects With Heart Failure Using Surgical Techniques Other Than Full Median Sternotomy
Brief Title: Implantation of the HeartMate 3 in Subjects With Heart Failure Using Surgical SWIFT HM3 PMS
Acronym: SWIFT
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10335VerC
Record Dates: First submitted 2020-06-19; First posted 2020-09-14 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Advanced Refractory Left Ventricular Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Treatment Arm: The treatment arm will have the HM3 LVAS implanted utilizing a technique other than full median sternotomy (e.g. thoracotomy).
  Interventions: Device: HeartMate 3 Left Ventricular Assist System (HM3 LVAS)

INTERVENTIONS:
Device: HeartMate 3 Left Ventricular Assist System (HM3 LVAS) — This clinical trial investigates implant of the HM3 LVAS by techniques other than full median sternotomy.

SUMMARY:
This is a prospective, post-market, multi-center, non-blinded, single arm study of the HeartMate 3 Left Ventricular Assist System (LVAS). The objective of this study is to evaluate the implantation of the HM3 utilizing techniques other than full median sternotomy (e.g. thoracotomy) and impact on post-implant length of stay.

ELIGIBILITY:
Inclusion Criteria

1. Subject or Legal Representative has provided written informed consent by signing the study Informed Consent Form (ICF)
2. Subject must be ≥ 18 years of age at the time of informed consent
3. Subject is receiving the HM3 as their first LVAD
4. Body surface area (BSA) ≥ 1.2m2
5. Subject is NYHA Class III with dyspnea upon mild physical activity or NYHA Class IV
6. LVEF ≤ 25%
7. Subject is:

   1. Inotrope dependent OR
   2. Has CI<2.2 L/min/m2, while not on inotropes and meets one of the following criteria:

      * On optimal medical management (OMM), based on current heart failure practice guidelines for at least 45 out of the last 60 days and is failing to respond to therapy
      * Advanced heart failure for at least 14 days AND dependent on intra-aortic balloon pump (IABP) for at least 7 days
8. Females of child bearing age must agree to use adequate contraception

Exclusion Criteria

1. Subject has a planned concomitant procedure at time of implant (e.g. valve repair, CABG, ASD repair, etc)
2. Subject has greater than mild aortic insufficiency
3. Physiologically significant (i.e. requires intervention) atrial septal defect
4. Subject has severe right heart failure (RHF) (refer to Appendix 2 for guidance)
5. Subject has planned Bi-VAD support prior to enrollment
6. Presence of mechanical aortic valve that will not be either converted to bioprosthesis or oversewn at the time of LVAD implant
7. Subject has ongoing mechanical circulatory support (MCS) at the time of LVAD surgery other than IABP
8. Subject has a history of any organ transplant
9. Positive pregnancy test
10. Etiology of heart failure (HF) due to or associated with uncorrected thyroid disease, obstructive cardiomyopathy, pericardial disease, amyloidosis or restrictive cardiomyopathy
11. Technical obstacles which pose an inordinately high surgical risk, in the judgment of the investigator
12. Platelet count < 100,000 x 103/L (< 100,000/ml)
13. Psychiatric disease/disorder, irreversible cognitive dysfunction or psychosocial issues that are likely to impair compliance with the study protocol and LVAS management
14. History of confirmed, untreated AAA > 5 cm in diameter within 6 months of enrollment
15. Presence of an active, uncontrolled infection
16. Intolerance to anticoagulant or antiplatelet therapies or any other peri/post-operative therapy the investigator will require based upon the subjects' health status
17. Presence of any one of the following risk factors for indications of severe end organ dysfunction or failure:

    1. An INR ≥ 2.0 not due to anticoagulation therapy
    2. Total bilirubin > 43 μmol/L (2.5 mg/dl) or biopsy-proven liver cirrhosis
    3. History of severe chronic obstructive pulmonary disease (COPD) defined by FEV1/FVC < 0.7, and FEV1 <50% predicted
    4. Fixed pulmonary hypertension with most recent PVR ≥ 8 Wood units that is unresponsive to pharmacologic intervention
    5. History of stroke within 90 days prior to enrollment, or a history of cerebrovascular disease with significant (> 80%) uncorrected carotid stenosis
    6. Serum creatinine ≥ 221 μmol/L (2.5 mg/dl) or the need for chronic renal replacement therapy
    7. Significant peripheral vascular disease (PVD) accompanied by rest pain or extremity ulceration
18. Pre-albumin < 150mg/liter (15 mg/dl) or albumin <30 g/liter (3g/dl) (if only one available); pre-albumin <150mg/liter (15 mg/dl) and albumin <30 g/liter (3 g/dl) (if both available)
19. Subject has known hypo- or hyper-coagulable states such as disseminated intravascular coagulation and heparin-induced thrombocytopenia
20. Participation in any other clinical investigation that is likely to confound study results or affect the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female subjects from the general heart failure population.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Proportion of patients surviving at 6 months free of debilitating stroke (Modified Rankin Score > 3), device malfunction requiring re-operation to replace or remove the device, or conversion of the implant surgical approach to open sternotomy. | 6 Months
  The composite primary endpoint of the study is survival at 6 months free of debilitating stroke (Modified Rankin Score > 3), device malfunction requiring re-operation to replace or remove the device, or conversion of the implant surgical approach to open sternotomy.

SECONDARY OUTCOMES:
Length of Stay | Initial hospital stay, approximately 3 weeks
  Mean length of hospital stay from implant to hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Sami Somo, PhD, Study Director — Abbott
Locations (32):
- United States (31):
  - Baptist Health Medical Center, Little Rock, Arkansas
  - Stanford University Medical Center, Palo Alto, California
  - University of Coloardo Hospital, Aurora, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Shands at the University of Florida, Gainesville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - St. Vincent Medical Group, Indianapolis, Indiana
  - Kansas University Medical Center, Kansas City, Kansas
  - Ochsner Medical Center, New Orleans, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Spectrum Health Butterworth Hospital, Grand Rapids, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - University of Minnesota Medical Center Fairview, Minneapolis, Minnesota
  - Barnes-Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Mount Sinai Hosptial, New York, New York
  - New York-Presbyterian/Columbia University Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical College of South Carolina, Charleston, South Carolina
  - Cardiothoracic & Vascular Surgeons, Austin, Texas
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Methodist Healthcare System of San Antonio, San Antonio, Texas
  - Sacred Heart Medical Center, Spokane, Washington
  - University of Wisconsin, Madison, Wisconsin
- Foothills Medical Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No